CLINICAL TRIAL: NCT07141134
Title: Turnova: The Clinical Efficacy, Manpower Reduction, and Cost-Effectiveness of Turn-Assist Alternating Pressure Air Mattresses for Pressure Injury Prevention in the ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202505127DIPD
Record Dates: First submitted 2025-08-12; First posted 2025-08-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Critical Care, Intensive Care; Nursing Workload; Cost Analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSFM + Manual Turning (Standard Care) (Active Comparator): ICU patients are placed on a high-specification foam mattress with scheduled manual repositioning per unit protocol (target every 2 hours using pillows). All other care follows unit protocols.
  Interventions: Device: HSFM; Other: Manual Turning (with pillows, per protocol)
- TAPAM (Turn-Assist Alternating Pressure Air Mattress with Positioning Pillows) (Experimental): ICU patients receive a turn-assist alternating pressure air mattress that integrates pressure redistribution with automated lateral turning at preset intervals with positioning pillows. The mattress is used continuously during the ICU stay. All other care follows unit protocols.
  Interventions: Device: TAPAM; Other: Positioning Pillows

INTERVENTIONS:
Device: TAPAM — Device: Turn-Assist Alternating Pressure Air Mattress (TAPAM) Automated lateral turning with pressure redistribution.
  Arms: TAPAM (Turn-Assist Alternating Pressure Air Mattress with Positioning Pillows)
Device: HSFM — Device: High-Specification Foam Mattress (HSFM) Standard ICU care support surface.
  Arms: HSFM + Manual Turning (Standard Care)
Other: Manual Turning (with pillows, per protocol) — Nurse-performed scheduled manual turning (target every 2 hours, with pillows).
  Arms: HSFM + Manual Turning (Standard Care)
Other: Positioning Pillows — Supplemental pillows used to support and maintain patient position.
  Arms: TAPAM (Turn-Assist Alternating Pressure Air Mattress with Positioning Pillows)

SUMMARY:
Pressure injuries are common in intensive care unit (ICU) patients who cannot reposition themselves. International guidelines recommend using support surfaces to redistribute pressure and regular turning to prevent these injuries. In Taiwan, high-specification foam mattresses (HSFM) with manual turning remain the standard, but frequent repositioning is labor-intensive and challenging in settings with limited nursing staff. The Turn-Assist Alternating Pressure Air Mattress (TAPAM) integrates pressure redistribution with automated lateral turning, potentially reducing nursing workload while maintaining preventive effectiveness. This study will compare TAPAM with HSFM plus manual turning in ICU patients, evaluating manpower requirements, time spent, perceived effort, and clinical outcomes. A cost-effectiveness and cost-benefit analysis will be conducted to assess the overall value of TAPAM for pressure injury prevention in high-risk ICU populations.

DETAILED DESCRIPTION:
This prospective comparative study will be conducted in the ICUs of a tertiary medical center in Taiwan. Adult patients at high risk for pressure injury and requiring assistance for repositioning will be enrolled and assigned to one of two interventions: (1) TAPAM, providing alternating pressure relief and programmed lateral turning, or (2) HSFM with manual repositioning according to standard ICU protocol.

Primary outcomes include manpower feasibility (number of staff required, time per turning) and clinical effectiveness (incidence of new pressure injuries). Secondary outcomes include economic indicators such as equipment costs, labor cost savings, and overall cost-effectiveness.

Economic evaluation will be performed from the hospital perspective, incorporating both direct costs (equipment, supplies, labor) and indirect savings from prevented injuries. Results will provide real-world evidence on whether TAPAM can improve care efficiency, reduce staff workload, and deliver cost-effective pressure injury prevention in high-dependency ICU settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) admitted to medical or surgical intensive care units (ICUs).
* Admission time between 08:00 and 23:00.
* Clinical condition requires ICU-level care.

Exclusion Criteria:

* Repeat ICU admission during the study period.
* Unstable spinal fracture.
* Receiving cervical or skeletal traction.
* Body weight >180 kg (exceeds mattress weight limit).
* Declines participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Manpower requirements for turning and positioning | Through ICU stay, up to 30 days (average per patient).
  Number of staff members required for each turning episode.
Time spent on turning and positioning | Through ICU stay, up to 30 days (average per patient).
  Duration (in minutes) from start to completion of each turning episode.
Perceived exertion of turning task | Through ICU stay, up to 30 days (average per patient).
  Nurses' subjective rating of physical effort required for each turning episode, measured using the Perceived Exertion Scale (PES);The scale ranges from 1 (no exertion at all) to 10 (maximal exertion). Higher scores indicate greater perceived exertion (worse outcome).

SECONDARY OUTCOMES:
Incidence of new pressure injuries | From ICU admission through ICU discharge (up to 30 days).
  Proportion of patients developing a new pressure injury (Stage 1-4) during ICU stay.
Pressure injury incidence density | From ICU admission through ICU discharge (up to 30 days).
  Number of new pressure injuries per 1,000 patient-days.
Pressure injury deterioration rate | From ICU admission through ICU discharge (up to 30 days).
  Proportion of existing pressure injuries that progress to a more severe stage during ICU stay.
Pressure injury deterioration density | From ICU admission through ICU discharge (up to 30 days).
  Number of deteriorated pressure injuries per 1,000 patient-days.
Economic evaluation: Total care costs | Through study completion, up to 30 days after ICU discharge.
  Total direct and indirect care costs during ICU stay, reported in U.S. dollars (USD).
Pressure injury-free days | From ICU admission through ICU discharge (up to 30 days).
  Number of days without a new pressure injury during ICU stay.
Economic evaluation:Labor costs | From ICU admission through ICU discharge (up to 30 days).
  Nursing and staff labor costs related to turning and positioning, reported in U.S. dollars (USD)
Economic evaluation:Equipment costs | Through study completion, up to 30 days after ICU discharge.
  Equipment-related costs (e.g., mattress and positioning aids), reported in U.S. dollars (USD).
Economic evaluation: Cost-effectiveness ratio | Through study completion, up to 30 days after ICU discharge.
  Incremental cost-effectiveness ratio comparing intervention and control groups.
Economic evaluation : Cost-benefit ratio | Through study completion, up to 30 days after ICU discharge
  Cost-benefit ratio comparing intervention and control groups.

OTHER OUTCOMES:
Nurse satisfaction with TAPAM | At 3 months after implementation of the intervention.
  Satisfaction scores covering ease of use, functionality, and perceived clinical effectiveness, measured via structured questionnaire using a 5-point Likert scale (range 1-5; higher scores indicate greater satisfaction).
Patient comfort and satisfaction with TAPAM | At ICU discharge (up to 30 days after ICU admission).
  Patient-reported comfort and satisfaction scores with the mattress, measured via structured questionnaire (or proxy report if the patient is unable to respond), using a 5-point Likert scale (range 1-5; higher scores indicate greater satisfaction).
Adverse events related to TAPAM | From device initiation through ICU discharge (up to 30 days).
  Incidence of events such as tube dislodgement, device malfunction, or electrical failure during use.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study results will be disseminated only in aggregate form through publications and conference presentations. The decision not to share IPD is based on data privacy considerations and institutional policy restrictions.